CLINICAL TRIAL: NCT02008838
Title: Effects of Synbiotic Supplementation in Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Assisstant Prof, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 450
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Synbiotic (Active Comparator): Each synbiotic capsule (Protexin, UK) contained 2 × 108 CFU of seven strains of friendly bacteria (Lactobacillus casei, Lactobacillus rhamnosus, Streptococcus thermophilus, Bifidobacterium breve, Lactobacillus acidophilus, Bifidobacterium longum, Lactobacillus bulgaricus), prebiotics (FOS [Fructooligosaccharide]), and probiotics culture (Magnesium stearate [source: mineral and vegetable], and vegetable capsule [hydroxypropyl methyl cellulose])
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): 250 mg Maltodexterin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic
  Arms: Synbiotic
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the effects of synbiotic supplementation on insulin resistance, and lipid profile in subjects with metabolic syndrome, in a randomized, double-blind, placebo-controlled pilot study, 38 subjects with metabolic syndrome will be supplemented with either synbiotic or placebo capsules twice/day for 28 weeks. Both the synbiotic (G1) and the placebo (G2) groups will be advised to follow an energy balanced diet and physical activity recommendations. Parameters related to metabolic syndrome and insulin resistance will be measured every 7 weeks during the study course.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* having three of the following five features: Increased waist circumference (≥102 cm in men and ≥88 cm in women), elevated TG (≥150 mg/dl), reduced HDL-C (≤40 mg/dl in men and ≤50 mg/dl in women), elevated blood pressure (≥130/85 mm Hg or on treatment for hypertension) and elevated glucose (≥100 mg/dl), according to the National Cholesterol Education Program Adult Treatment Panel III report
* BMI : 25≥ BMI ≥ 40

Exclusion Criteria:

* Use antibiotic 2 weeks before recruitment to the study
* A history of alcohol consumption
* Pregnancy & Breast feeding , Professional athelets
* A history of Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 28 weeks